CLINICAL TRIAL: NCT06301243
Title: Molecular Signature of Inactivity Induced Exercise Responsiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University Wisconsin (Other)
Responsible Party: Principal Investigator, Kevin Gries, Assistant Professor, Concordia University Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FY24-62
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Diseases; Aerobic Exercise
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inactive (Experimental): Subjects will be asked to be sedentary prior to an acute exercise bout (<5,000 steps as measured by a physical activity monitor).
  Interventions: Other: Inactivity
- Normal activity (Placebo Comparator): Subjects will be asked to have normal activity prior to an acute exercise bout (>8,500 steps as measured by a physical activity monitor).
  Interventions: Other: Inactivity

INTERVENTIONS:
Other: Inactivity — Low physical activity level prior to the exercise intervention.
  Other Names: Sedentary

SUMMARY:
Fitness is one of the best predictors for heart and brain disease. To increase ones fitness, the American Heart Association (AHA) says to exercise at least 150 minutes per week or 75 minutes per week if really hard. These exercise guides are pretty effective, however not everyone will get the same results. What individuals do outside of the exercise bout can influence the effectiveness of exercise. One of these factors is our time sitting, which has caused the phrase "sitting is the new smoking". Other studies have said that the metabolic benefits of exercise are decreased when you exercise after a few days of low activity (less than 5,000 steps per day). This is important in that exercise may not be able to fully offset these times of inactivity. However, these studies were only looking at different fats in the blood. As exercise increases fat burn up to 10 times in the muscle, more research is needed to understand how inactivity affects the muscle during exercise and after exercise. This study will help answer two questions: 1) How does a day of sitting a lot affect the muscle's ability to respond to exercise? and 2) How does a day of sitting a lot affect carbohydrate and fat burn during and after a bout of exercise? The investigators will answer these questions by having people complete one day of inactivity (less than 5,000 steps) or normal activity (more than 8,500 steps). Subjects will then come in the next day to bike somewhat hard for 1 hour. The investigators will take blood samples before, during, and after exercise to measure energy sources. The investigators will also collect pieces of skeletal muscle before and after exercise to see how the muscle responded to exercise. This study is significant for the publication of exercise guidelines to minimize risk of heart and metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* free from acute or chronic illness (cardiac, pulmonary, liver, or kidney abnormalities, cancer, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other known metabolic disorders)
* free from orthopedic limitations (including any artificial joints) no known lidocaine allergy
* do not currently smoke or participate in other forms of tobacco use.
* not currently in a structured exercise program

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Circulating lipid and carbohydrate metabolism | Baseline; 20 and 40, and 60 minutes into exercise; and every 30 minutes after exercise up to 4 hours
  Investigate the role of sex and inactivity on lipid and carbohydrate metabolism following a bout of aerobic exercise.
Basal and post-exercise gene expression with inactivity | Baseline; 4 hours after exercise
  Study the role of inactivity on basal and exercise-induced gene expression in skeletal muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Kevin J Gries, Mequon, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes